CLINICAL TRIAL: NCT00000434
Title: Impact of Exercise on Older Persons With Osteoarthritis (OA)
Brief Title: Impact of Exercise on Older Persons With Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Susan Hughes, Center for Research on Health and Aging, UIC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P60AR030692 (NIH); NIAMS-050
Record Dates: First submitted 2000-01-21; First posted 2000-01-24 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2007-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Health education; Aerobic exercise; Self-efficacy; Muscle strength; Outcomes research; Longitudinal study
MeSH Terms: conditions — Osteoarthritis; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Fit and Strong! is a multi-component exercise and health education program that incorporates flexibility, aerobic conditioning, strength training, and group discussion/problem solving for lifestyle change.
  Interventions: Behavioral: Fit and Strong!

INTERVENTIONS:
Behavioral: Fit and Strong! — Fit and Strong! is a multi-component exercise and health education program that includes flexibility, aerobic conditioning, strength training, and group discussion/problem solving for lifestyle change.

SUMMARY:
Previous studies have found that exercise can reduce pain, improve endurance for physical activities, and improve cardiovascular fitness over time. However, these studies have not looked at the impact of exercise programs for older adults with osteoarthritis or at how long older adults continue exercising after a program is finished. This study will look at the long-term effects of a structured exercise program for people aged 60 or older who have osteoarthritis of the hip or knee. One goal of the exercise program is to encourage older people with osteoarthritis to continue exercising.

We will randomly assign study participants to either the exercise program or a control group that does not do the exercise program. We will monitor participants at the start of the study, at 8 weeks, and every 3 months for 2 years after the program is completed. The exercise program lasts for 8 weeks and includes an exercise part and an educational part led by trained physical therapists. We believe that participants in the treatment (exercise) group will show higher rates of continued exercise and higher functional status over time compared to the group of people who do not participate in the exercise program.

DETAILED DESCRIPTION:
Recent exercise interventions have demonstrated statistically significant short-term improvements in muscle strength, fitness, and physical activity in people under the age of 70. This study seeks to determine if those same benefits can be achieved in an older population (mean age 84) with osteoarthritis of the hip or knee. The study will examine the long-term effects of a structured exercise program that seeks to promote adherence to continued exercise.

We will randomly assign people who meet the study criteria to the exercise intervention or control group. We will conduct measures at baseline, at 8 weeks, and at 3-month intervals for 2 years following the intervention. The exercise component of the intervention will include lower extremity muscle strengthening, range-of-motion exercises, and fitness walking. An educational component will focus on arthritis self-efficacy and perceived self-reported exercise efficacy. We hypothesize that treatment group participants will exhibit higher rates of adherence to exercise and higher functional status outcomes over time compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Presence of osteoarthritis of the lower extremities with an American College of Rheumatology functional class rating of I, II, or III
* No other contraindication from a personal physician for participation in the fitness walking
* Lack of moderate-to-severe cognitive impairment as assessed by the Short Portable Mental Status Questionnaire

Exclusion Criteria:

* Under 60 years of age
* Lack of osteoarthritis of the lower extremities
* Contraindication from a personal physician for participation in fitness walking
* Presence of moderate-to-severe cognitive impairment as assessed by the Short Portable Mental Status Questionnaire
* Steroid injections in either hip or knee within the previous 6 months
* Uncomplicated knee or hip surgery within previous year
* Complicated knee or hip surgery within previous year
* Plans for total knee or hip replacement within the next year
* Rheumatoid arthritis or other systemic inflammatory arthritis
* Diabetes that is not under control
* Current participation in a structured aerobic exercise program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 1983-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Adherence to exercise | 12 months

SECONDARY OUTCOMES:
Pain and stiffness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hughes, Principal Investigator — Center for Research on Health and Aging
Locations (2):
- United States (2):
  - North Park Village, Chicago, Illinois
  - Bernard Horwich Jewish Community Center, Chicago, Illinois

REFERENCES:
- [Background] Hughes SL, Seymour RB, Campbell R, Pollak N, Huber G, Sharma L. Impact of the fit and strong intervention on older adults with osteoarthritis. Gerontologist. 2004 Apr;44(2):217-28. doi: 10.1093/geront/44.2.217. PMID 15075418
- [Background] Hughes SL, Seymour RB, Campbell RT, Huber G, Pollak N, Sharma L, Desai P. Long-term impact of Fit and Strong! on older adults with osteoarthritis. Gerontologist. 2006 Dec;46(6):801-14. doi: 10.1093/geront/46.6.801. PMID 17169935